CLINICAL TRIAL: NCT06185101
Title: A Feasibility Study of a Chronic Pain Self-management Intervention for Older Adults Incorporating Podcasts and Patient Priorities
Brief Title: Support, Training, and Education for Pain Self-Management Using Podcasts: A Pilot Trial
Acronym: STEP-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Western Wayne Family Health Centers (Unknown); National Institute on Aging (NIA) (NIH); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary Janevic, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00240183; 5P30AG022845-20 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Palliative Care; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEP-UP intervention group (Experimental): Participants will engage in a behavioral intervention for pain self-management that incorporates educational podcasts and sessions with a community health worker.
  Interventions: Behavioral: STEP-UP
- Control group (No Intervention): Members of the control group will not initially receive the STEP-UP intervention. After completing the 8-week follow-up telephone survey, individuals in the control group will be invited to take part in the STEP-UP intervention.

INTERVENTIONS:
Behavioral: STEP-UP — The STEP-UP chronic pain self-management intervention (Support, Training, and Education for Pain Self-Management - Using Podcasts) will feature an educational podcast series teaching core pain self-management skills. Podcasts will be supplemented by sessions with a Community Health Worker taking place at designated times over a 7-week period. The Community Health Worker will guide participants in a modified Patient Priorities of Care (PPC) approach to help them identify their values and priorities and develop goals that reflect these.
  Other Names: Support, Training, and Education for Pain self-management, Using Podcasts
  Arms: STEP-UP intervention group

SUMMARY:
This randomized Stage 1 pilot trial tests the feasibility of a community health worker (CHW) delivered chronic pain self-management intervention for older adults ("STEP-UP"; Support, Training, and Education for Pain Self-Management - Using Podcasts) in a primary care setting. A total of 40 participants aged 50+ with high-impact chronic pain will be randomized to intervention or control groups. The STEP-UP intervention will feature an educational podcast series teaching core pain self-management skills. Podcasts will be supplemented by sessions with a Community Health Worker taking place at designated times over a 7-week period. The Community Health Worker will guide participants in a modified Patient Priorities of Care approach to help them identify their values and priorities and develop goals that reflect these.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Have a mobile or landline phone
* Report high-impact chronic musculoskeletal pain (defined as pain in muscles or joints for > 3 months "most days" or "every day" on a scale of never, some days, most days, or every day) AND their pain limited life or work activities over the past 3 months "most days" or "every day"
* Have not participated in another chronic pain self-management intervention in the last 5 years.
* Able to converse comfortably in English

Exclusion Criteria:

* Serious acute illness or hospitalization in the last month;
* Planned major surgery in the next three months that would interfere with program participation (e.g., knee or hip replacement)
* Severe cognitive impairment or other severe physical or psychiatric disorder judged by the study team to pose a significant barrier to participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STEP-UP Intervention Group | Control Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STEP-UP Intervention Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.85 (5.81) | 58.3 (6.12) | 59.08 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Interference 6-item Subscale From PROMIS-43 Adult Profile
Description: Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much); raw total scale scores range from 6 (low interference) to 30 (high interference). Scores are converted to a standardized T-score metric, with a mean of 50 and a standard deviation of 10 in a referent population. A higher score means more of the concept being measured. Change scores are calculated as [8 week score] - [baseline score]; therefore, a greater negative value means a greater reduction in pain interference.
Time Frame: Baseline, 8 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
score on a scale | -3.3 (7.8) | -3.7 (8.2)
Statistical Analysis 1: Comparison: STEP-UP Intervention Group vs Control Group; Test type: Superiority; p = 0.84, Regression, Linear; Adjusted for age and gender

2. Secondary Outcome: Global Impression of Change in Pain
Description: How participant thinks their pain has changed from baseline (much worse (-3) to much better(+3)).
Time Frame: 8 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
score on a scale | 0.9 (1.07) | 0.25 (1.45)

3. Secondary Outcome: Global Impression of Change in Functioning
Description: How participant thinks their functioning has changed from baseline (much worse (-3) to much better(+3)).
Time Frame: 8 weeks from baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP Intervention Group | Control Group
Number analyzed (Participants) | 20 | 20
score on a scale | 1.05 (0.89) | 0.5 (1.28)

4. Secondary Outcome: Engagement as Measured by Number of Sessions Completed
Description: Number of sessions out of 6 completed 8 weeks from baseline
Time Frame: 8 weeks from baseline
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | STEP-UP Intervention Group
Number analyzed (Participants) | 20
sessions | 5.2 (1.93)

5. Secondary Outcome: Participant Satisfaction
Description: Items ask about overall satisfaction with the program, e.g., whether participation increased understanding of pain management (1= Strongly Disagree to 5= Strongly Agree). A higher score indicates higher patient satisfaction.
Time Frame: 8 weeks from baseline
Population: Participants who attended any intervention sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-UP Intervention Group
Number analyzed (Participants) | 18
score on a scale | 4.33 (0.59)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | STEP-UP Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEP-UP Intervention Group (N=20) | Control Group (N=20)
hospitalization (Cardiac disorders) | 1 (1) | 0
hospitalization (Infections and infestations) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEP-UP Intervention Group (N=20) | Control Group (N=20)
unexplained bleeding (General disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT06185101/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT06185101/ICF_001.pdf